CLINICAL TRIAL: NCT04271319
Title: Efficacy of a High Voltage Pulsed Current in the Non-Invasive Treatment of Carpal Tunnel Syndrome
Brief Title: Avazzia HVPC Bio-Electrical Stimulation Technology (BEST™) Microcurrent CTS RCT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Avazzia, Inc (Industry)
Collaborators: Joseph Surace, D.C. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: RA-190930-CTS-01
Record Dates: First submitted 2020-01-22; First posted 2020-02-17 (Actual); Last update posted 2021-07-27 (Actual); Status verified 2021-07

CONDITIONS: Carpal Tunnel Syndrome
Keywords: musculoskeletal disorder; median nerve; carpal tunnel; hand numbness; electric stimulation; microcurrent
MeSH Terms: conditions — Carpal Tunnel Syndrome; Musculoskeletal Diseases; Median Neuropathy

STUDY DESIGN:
Intervention Model Description: Device: Avazzia Pro-Sport Ultra® device
  High-voltage pulsed current (HVPC) electrical stimulation with Reactions and BEST™ (Bio-Electric Stimulation Technology) microcurrent that measure and change with tissue electrical characteristics.
Who Masked: Participant, Investigator
Masking Description: Double (participant, care provider)
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- BEST™ Pro-Sport Ultra® microcurrent device (Experimental): Participants will receive treatment with an active electrical stimulation device for 7 in-clinic treatments over 2 weeks.
  Interventions: Device: BEST™ HVPC microcurrent electrical stimulation PRO-SPORT Ultra® Device
- Electrical Stimulation - Sham Comparator (Sham Comparator): Participants will receive treatment with a sham electrical stimulation device for 7 in-clinic treatments over 2 weeks.
  Interventions: Device: Sham PRO-SPORT Ultra® Device

INTERVENTIONS:
Device: BEST™ HVPC microcurrent electrical stimulation PRO-SPORT Ultra® Device — Participants will receive treatment with an active electrical stimulation device for 7 in-clinic treatments over 2 weeks.
  Active Avazzia PRO-Sport Ultra® medical device, BEST™ HVPC microcurrent electrical stimulation, FDA cleared for pain relief
  Arms: BEST™ Pro-Sport Ultra® microcurrent device
Device: Sham PRO-SPORT Ultra® Device — Participants will receive treatment with a sham electrical stimulation device for 7 in-clinic treatments over 2 weeks.
  Sham PRO-SPORT Ultra® device will be used. The built in electrodes and the accessory port for connecting the lead wire to the electrode pads will be disconnected internal to the device. The device will power on with the same sounds and indications.
  Arms: Electrical Stimulation - Sham Comparator

SUMMARY:
A clinical study at Activated Family Chiropractic & Wellness, is being proposed to test the efficacy of a novel electrical stimulation platform named the Pro-Sport Ultra® designed by AVAZZIA to relieve pain and improve mobility in patients with Carpal Tunnel Syndrome (CTS).

DETAILED DESCRIPTION:
This study will recruit patients with a prior diagnosis (Dx) of CTS and have had a trial of conservative treatment for a minimum of 4 weeks without successful results due to continuing symptoms that interfere with normal function.

The primary objective of this study is to compare the changes obtained in CTS that have not successfully responded to non-surgical management by incorporating PRO-Sport Ultra® as opposed to an inactive device. This study aims to compare improvement obtained in CTS using the new therapy.

All participants will be randomized into two treatment groups and receive treatment with both active and inactive devices during the study. During the first 2 weeks, one group will receive treatment with the active device and the other group will receive treatment with the inactive device. At the end of week 3 (no treatment week), participants will return to the clinic and will be crossed over for the next 2 weeks of treatment.

The Avazzia PRO-Sport Ultra® and BEST-RSI® devices are non-invasive, hand-held, battery operated microcurrent devices that are FDA-cleared for the symptomatic relief and management of chronic, intractable pain and adjunctive treatment in the management of post-surgical and post-traumatic pain.

ELIGIBILITY:
Inclusion Criteria:

* Have a prior diagnosis (Dx) of CTS and have had a trial of conservative treatment for a minimum of 4 weeks without successful results due to continuing symptoms that interfere with normal function.
* Confirmation of this Dx shall include at least three findings as defined below:

  * Muscle atrophy, severe weakness of thenar muscles
  * 2-point discrimination test >6mm
  * Flick sign (shaking hand)
  * Phalen's sign
  * Tinel's sign
  * Reverse Phalen's sign
  * Abnormal Katz hand diagram scores
  * Positive NCV testing
* Age >18 - <70 years old
* Males/Females of all ethnicities
* Post-surgical failures >6 months post op
* Ability to understand the informed consent document before signing it

Exclusion Criteria:

* Systemic disease that would affect treatment outcome such as inflammatory joint diseases (i.e., rheumatoid arthritis, systemic lupus); malignancies undergoing treatment or any malignancies (in remission or not) with involvement of the musculoskeletal system.
* Co-morbidities, thoracic outlet nerve impingement, neuropathy, etc. should be identified and, if significant, the candidate should be excluded from the study.
* Cubital tunnel syndrome, anterior and posterior interosseous nerve syndrome, lateral and medial epicondylitis, handlebar palsy, De Quervain's disease, trigger finger, and Intersection syndrome should be differentiated from CTS and not included in this study.
* Uncontrolled mood disorders, such as depression, anxiety.
* Drug or substance abuse within past 90 days.
* Any hand pathology requiring surgical intervention.
* Active litigation, workers compensation
* Any participant with an electrically implanted device such as a pacemaker, neural stimulator, etc.
* Participant is currently pregnant, nursing, or may become pregnant.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-09-14 (Actual); Primary Completion 2021-08-31 (Estimated); Study Completion 2021-08-31 (Estimated)

PRIMARY OUTCOMES:
Pain Level Assessment | 5 weeks
  Change in pain associated with CTS during visit #1, 7, 8 ,14, and visit 15 [Time Frame: baseline to 5 weeks] Pain will be assessed with VAS (Visual Analog Scale pain score) from 0 to 10 where 10 is the worst pain ever.
Motor Function Examination | 5 weeks
  Change in the score of motor function examination during visit #1, 7, 8 ,14, and visit 15 [Time Frame: baseline to 5 weeks] Change will be assessed using the motor function score from 0 to 5 where 5 is full range of motion.
Nerve Conduction Velocity | 5 weeks
  Nerve conduction velocity during visit #1, 7, 8 ,14, and visit 15 [Time Frame: baseline to 5 weeks] Change in nerve conduction velocity will be assessed from the score obtained from testing done by the Mediracer Carpal Tunnel Syndrome Sensory exam from normal to severe.

SECONDARY OUTCOMES:
Healthy Related Quality of Life Changes | 5 weeks
  Change in health Related Quality of Life during visit #1, 7, 8 ,14, and visit 15 [Time Frame: baseline to 5 weeks] Change will be assessed with QuickDash score from 0 to 100 where 100 is most severe disability.
Sensory ability changes | 5 weeks
  Change in sensory ability during visit #1 and 15 [Time Frame: baseline to 5 weeks] Change will be assessed with Katz Hand Diagram.
Dosage/Frequency of Analgesics changes | 5 weeks
  Change in frequency and dosage of analgesics during visit #1, 7, 8 ,14, and visit 15 [Time Frame: baseline to 5 weeks] Change will be assessed with comparison of frequency and analgesics from visit to visit.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Surace, D.C., Principal Investigator — Activated Family Chiropractic & Wellness
Locations (1):
- Activated Family Chiropractic and Wellness, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: No